CLINICAL TRIAL: NCT03689179
Title: Virtual Coaching to Maximize Dementia Caregivers' Respite Time-Use: A Stage 1 Pilot Test for Feasibility and Efficacy
Brief Title: Virtual Coaching to Maximize Dementia Caregivers' Respite Time Use
Acronym: TLC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Rebecca Utz, Associate Professor, University of Utah
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 1R01AG061946-01 (Utz); R01AG061946 (NIH)
Record Dates: First submitted 2018-09-19; First posted 2018-09-28 (Actual); Results first posted 2024-03-05 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Anxiety; Burden, Dependency; Caregiver
MeSH Terms: conditions — Anxiety Disorders | interventions — Time

STUDY DESIGN:
Intervention Model Description: This study uses a full-powered pilot sample (n=150) and a randomized waitlist control design to examine feasibility and initial efficacy of the TLC intervention. After an initial orientation/control period (4 weeks), group A will receive access to the TLC intervention for 8 weeks, followed by an optional 8-week control period where they can continue to use the TLC intervention if they choose. After the initial 4-week orientation period, Group B will receive 8 weeks of waitlist (no treatment) control, followed by access to the TLC intervention for 8 weeks. Primary outcomes (defined as anxiety, caregiver burden) will be assessed by electronically delivered surveys every 4 weeks; respite time-use and time-use satisfaction will be assessed using ecological momentary analysis for each respite period taken during the 20-week study period; feasibility will be assessed using fixed-choice and open-ended survey questions collected post-intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment with Follow-up (Group A) (Experimental): Group A received access to the full "Time for Living & Caring" (TLC) intervention for 8 weeks (calendar + coaching + resources), followed by an 8-week maintenance period where they could continue to use the TLC intervention. The TLC intervention turned off after 16 weeks of exposure for all participants.
  Interventions: Behavioral: Time for Living and Caring (TLC)
- Wait-List Control w/Treatment (Group B) (Experimental): Group B received 8 weeks of waitlist control (minimal treatment - calendar only) , followed by access to the full "Time for Living & Caring" (TLC) intervention for an additional 8 weeks (calendar + coaching + resources). The TLC intervention turned off after 16 weeks of exposure for all participants.
  Interventions: Behavioral: Time for Living and Caring (TLC)

INTERVENTIONS:
Behavioral: Time for Living and Caring (TLC) — "Time for Living & Caring" (TLC) is an online, self-administered intervention. It includes three types of modules: 1) "virtual coaching" module (defined as a series of prompts, reminders, and suggestions that guide caregivers through assessment, goal setting, and goal review activities) to monitor respite time-use and time-use goals, 2) an interactive calendar that can be used to schedule and track respite time, 3) resource pages (including links, printable forms, video guides) that provide education and resources such as What is Respite?, Why is Respite Important?, How do I Get (More) Respite?, How do I Use Respite?.

SUMMARY:
The "Time for Living & Caring" (TLC) intervention is an online, self-administered intervention, with the purpose of providing informal family caregivers with resources, support, and education to maximize the benefit of their respite time-use (respite is defined as planned time away from caregiving; it can be provided by a formal service provider or informal arrangements within families/networks). The study will use a full-powered pilot sample (anticipated n=150; actual n=166) and a randomized waitlist control design to examine feasibility and initial efficacy of the TLC intervention.

DETAILED DESCRIPTION:
The purpose of this study is to redevelop the Time for Living and Caring (TLC) intervention, in which dementia caregivers are taught strategies to assess and identify ways to spend upcoming periods of respite time, to a fully online, self-administered virtual coaching format, and then to pilot-test the new TLC intervention for feasibility and efficacy.

Aim 1 is to modify, adapt, and refine the existing intervention modules, utilizing a community-engaged design process where stakeholders (i.e., current or former caregivers, diverse community leaders, and respite providers) will work as consultants alongside the research, technical, and creative teams to develop and provide feedback on the TLC prototypes. The primary endpoint of this phase of the study is a fully-developed, tested, and ready-to-launch web-based intervention.

Aim 2 is to conduct a pilot test with dementia caregivers who are currently using respite, using a full powered pilot sample and a randomized waitlist-control experimental design where participants are exposed to the redeveloped TLC intervention for 8 weeks and will provide assessments of daily respite use, respite time-use satisfaction, and wellbeing. These pilot data will be used to assess feasibility and to explore hypotheses regarding the potential efficacy of the intervention as well as the mechanism - time-use satisfaction -underlying the intervention's effect on wellbeing. **Aim 2 uses a clinical trial methodology, and is therefore the part of the study that is described in detail here **

Aim 3 is intended to explore future implementation with respite providers, as yet another assessment of the intervention's feasibility. We will host webinars to demonstrate the features and functionality of the TLC intervention. We will then ask providers for feedback on their likelihood of implementation and barriers to using TLC with their clients.

Together, these three aims represent a comprehensive approach to Stage 1 behavioral intervention research activities, with the overall goal of (re)developing an intervention that is useful to dementia caregivers and is scalable to real world applications. Each aim has a separate sample and study design.

Aim 1 Sample & Design: a dozen community stakeholders, consisting of current and former AD/ADRD caregivers, respite providers, and community leaders that represent diverse local populations. These participants will be considered "consultants" (not human subjects), per IRB. They are providing feedback and advice to the research team and technical designers in the creation and translation of the TLC intervention tools to a self-administered, app-delivered intervention.

Aim 2 Sample & Design: a total of 150 respite-using AD/ADRD caregivers. This is the sample that is participating in the clinical trial. ** eligibility, measures, study design for this phase of the overall project are described in greater detail here **

Aim 3 Sample & Design: a minimum of 100 respite providers, located anywhere in the US, such as staff from home health agencies, adult day care centers, area agencies on aging, long term care communities, hospices, hospitals, etc. Eligibility is based on their interest and willingness to learn more about the TLC intervention. This sample will provide feedback on the features and functionality of the TLC intervention, as well as specific advice on how it could serve their clients and be disseminated in the future. This is human subjects research, but is not part of the clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* caregivers to persons with Alzheimer's Disease or Related Dementia (AD/ADRD) (self-identified)
* use formal or informal respite for at least 4 hours per week.
* primary caregiver (self-identified)
* co-residing with the care recipient
* 18 years or older AND
* able to read and write in English.

Exclusion Criteria:

* caregivers to persons with disability or chronic condition, and not Alzheimer's Disease and Related Dementia (AD/ADRD)
* caregivers who do not use respite for at least 4 hours per week
* noncoresidential caregivers
* younger than 18 years
* not able to read and write in English

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2020-10-20 (Actual); Primary Completion 2022-08-05 (Actual); Study Completion 2024-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: rebecca utz, PhD, Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared with investigators working under an institution with a Federal Wide Assurance (FWA) and can be used for secondary data analyses by investigators outside of the original TLC study team. The PI agrees to make available data within one year of the completion of the funded project period. De-identified individual data will be available directly from the PI. The PI agrees to share data and resources in a manner that is fully consistent with NIH data and resource sharing policies and applicable laws and regulations.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Within one year of the completion of the funded project period.
Access Criteria: Investigators working under an institution with a Federal Wide Assurance (FWA) can email the PI directly, asking for permission

REFERENCES:
- [Derived] Iacob E, Caserta M, Donaldson G, Sparks C, Terrill A, Thompson A, Wong B, Utz RL. Evaluating the Efficacy of Time for Living and Caring: An Online Intervention to Support Dementia Caregivers' Use of Respite. Innov Aging. 2024 Apr 26;8(5):igae043. doi: 10.1093/geroni/igae043. eCollection 2024. PMID 38803611

RESULTS

PARTICIPANT FLOW:
Groups:
- Wait-List Control (Group B): Group B received 8 weeks of waitlist control (minimal treatment - calendar only) , followed by access to the full "Time for Living & Caring" (TLC) intervention for an additional 8 weeks (calendar + coaching + resources). The TLC intervention turned off after 16 weeks of exposure for all participants.
  Time for Living and Caring (TLC): "Time for Living & Caring" (TLC) is an online, self-administered intervention. It includes three types of modules: a "virtual coaching" module (defined as a series or prompts, reminders, and suggestions delivered electronically through an interactive calendar website) that guides caregivers through assessment, goal setting, and goal review activities using an interactive calendar for each planned respite period they have. Supplementary modules provide education and resources such as What is Respite?, Why is Respite Important?, How do I Get (More) Respite?, How do I Use Respite?.
Period: Overall Study
Arm/Group | Treatment With Follow-up (Group A) | Wait-List Control (Group B)
Started | 83 | 83
Completed | 69 | 67
Not Completed | 14 | 16

BASELINE CHARACTERISTICS:
Groups:
- Waitlist Control (Group A): Group B received 8 weeks of waitlist control (minimal treatment - calendar only) , followed by access to the full "Time for Living & Caring" (TLC) intervention for an additional 8 weeks (calendar + coaching + resources). The TLC intervention turned off after 16 weeks of exposure for all participants.
- Total: Total of all reporting groups
Arm/Group | Treatment With Follow-up (Group A) | Waitlist Control (Group A) | Total
Number analyzed (Participants) | 83 | 83 | 166
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.8 (13.1) | 62.6 (12.9) | 61.7 (13.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 66 | 65 | 131
  Male | 17 | 18 | 35
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 2 | 9
  Not Hispanic or Latino | 76 | 74 | 150
  Unknown or Not Reported | 0 | 7 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 1 | 3 | 4
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 4 | 5 | 9
  White | 71 | 66 | 137
  More than one race | 4 | 1 | 5
  Unknown or Not Reported | 0 | 8 | 8
Region of Enrollment [Number; unit: participants]
  United States | 83 | 83 | 166
Marital Status [Count of Participants; unit: Participants]
  Married | 65 | 69 | 134
  Divorced | 8 | 4 | 12
  Living with Partner | 3 | 2 | 5
  Never Married | 5 | 2 | 7
  Widowed | 2 | 0 | 2
  Unknown or Not Reported | 0 | 6 | 6
Education Completed [Count of Participants; unit: Participants]
  Some High School | 2 | 1 | 3
  High School Graduate | 4 | 4 | 8
  Some College, Associates Degree, and/or Vocational or Technical School | 33 | 27 | 60
  College or University Degree | 22 | 24 | 46
  Postgraduate or Professional Degree | 21 | 22 | 43
  Unknown or Not Reported | 1 | 5 | 6
Annual Income [Count of Participants; unit: Participants]
  $10,000 to $19,999 | 2 | 0 | 2
  $20,000 to $29,999 | 6 | 7 | 13
  $30,000 to $39,999 | 7 | 1 | 8
  $40,000 to $49,999 | 8 | 8 | 16
  $50,000 to $59,999 | 10 | 12 | 22
  $60,000 to $69,999 | 12 | 8 | 20
  $70,000 to $79,999 | 3 | 8 | 11
  $80,000 to $89,999 | 5 | 6 | 11
  $90,000 to $99,999 | 7 | 4 | 11
  $100,000 to $149,999 | 17 | 11 | 28
  $150,000 or more | 4 | 13 | 17
  Unknown or Not Reported | 2 | 5 | 7

OUTCOME MEASURES:

1. Primary Outcome: Anxiety Symptoms, as Measured by PROMIS Anxiety Short Form
Description: Anxiety was measured with the PROMIS Anxiety short-form questionnaire for adults, a self-report, 8-item additive scale that standardizes the distribution of anxiety-related symptoms (T-score) on a population-distribution with a mean of 50 and standard deviation of 10: "During the past 7 days, I felt nervous, anxious, fearful, uneasy, tense, worried, unable to focus on anything other than my anxiety, felt like I needed help with my anxiety" each assessed with a five-category response (never, rarely, sometimes, often, always). Higher scores indicate a higher level of anxiety.
Time Frame: Baseline (week 1, pre-intervention), week 4, week 8, week 12, week 16 (post-intervention) and week 20 (follow-up) for both Group A and Group B
Population: Three enrolled participants were excluded from this analysis due to missing baseline data (i.e., 163 person out of 166 enrolled have data).If a participant was missing more than 30% of the items (i.e., 2 or more items on the anxiety questionnaire), the scale score was coded as missing. Under these criteria, the full TLC sample has a calculated score for anxiety.
Measure: Mean (95% Confidence Interval); unit: T-score
Groups:
- Treatment With Follow-up (Group A): Group A will receive access to the full "Time for Living & Caring" (TLC) intervention for 16 weeks, with a 4-week follow-up at Week 20 of the study.
  Time for Living and Caring (TLC): "Time for Living & Caring" (TLC) is an online, self-administered intervention. It includes three types of modules: a "virtual coaching" module (defined as a series or prompts, reminders, and suggestions delivered electronically through an interactive calendar website) that guides caregivers through assessment, goal setting, and goal review activities using an interactive calendar for each planned respite period they have. Supplementary modules provide education and resources such as What is Respite?, Why is Respite Important?, How do I Get (More) Respite?, How do I Use Respite?.
- Wait-List / Control Treatment With Follow-up (Group B): After the initial 8-week orientation period where Group B will receive 8 weeks of waitlist (limited treatment) control, followed by full access to the "Time for Living & Caring" (TLC) intervention for 8 weeks. They will also receive a 4-week follow-up at Week 20 of the study.
  Time for Living and Caring (TLC): "Time for Living & Caring" (TLC) is an online, self-administered intervention. It includes three types of modules: a "virtual coaching" module (defined as a series or prompts, reminders, and suggestions delivered electronically through an interactive calendar website) that guides caregivers through assessment, goal setting, and goal review activities using an interactive calendar for each planned respite period they have. Supplementary modules provide education and resources such as What is Respite?, Why is Respite Important?, How do I Get (More) Respite?, How do I Use Respite?.
Arm/Group | Treatment With Follow-up (Group A) | Wait-List / Control Treatment With Follow-up (Group B)
Number analyzed (Participants) | 83 | 80
T-score
  T0 - baseline, Pre-Intervention | 55.51 [53.48 to 57.53] | 53.93 [51.95 to 55.90]
  T4 | 56.75 [54.65 to 58.86] | 57.35 [55.50 to 59.21]
  T8 | 56.39 [54.38 to 58.40] | 56.99 [55.38 to 58.59]
  T12 | 56.92 [54.76 to 59.09] | 54.20 [52.53 to 55.86]
  T16 - Post Intervention | 56.54 [54.24 to 58.85] | 52.75 [50.75 to 54.75]
  T20 - Follow-up | 58.15 [55.79 to 60.52] | 55.73 [53.69 to 57.77]

2. Primary Outcome: Caregiver Burden Score, as Measured by "Caregiver Burden Inventory"
Description: Self-report multi-item index (24 items; range 0-96). Lower scores indicate lower levels of caregiver burden. Higher scores indicate higher levels of perceived burden associated with caregiving tasks.
Time Frame: as for outcome 1
Population: Three enrolled participants were excluded from analysis due to missing baseline data.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Treatment With Follow-up (Group A) | Wait-List / Control Treatment With Follow-up (Group B)
Number analyzed (Participants) | 83 | 80
score on a scale
  T0 - Baseline | 45.94 [42.22 to 49.65] | 46.10 [42.40 to 49.79]
  T4 | 45.33 [41.39 to 49.27] | 43.22 [40.50 to 45.95]
  T8 - mid intervention | 45.02 [41.37 to 48.66] | 43.37 [40.16 to 46.58]
  T12 | 45.72 [41.66 to 49.78] | 40.80 [37.65 to 43.94]
  T16 - Post intervention | 49.91 [45.57 to 54.26] | 42.05 [38.31 to 45.79]
  T20 - follow up | 50.09 [45.47 to 54.71] | 43.23 [40.01 to 46.46]

3. Secondary Outcome: Respite Time-Use (in Hours Per Week)
Description: Participants were asked to self-report number of hours they typically receive respite in a typical week. The following survey question and description were asked to all participants "On average, how many hours of respite do you get in a typical week? These would be hours that you can completely turn-off your caregiving responsibilities, while the needs and safety of your family member are not your primary responsibility."
Time Frame: Pre-Intervention (baseline, week 1) and Post-Intervention (week-16) for both Group A and Group B
Population: Three enrolled participants were excluded from this analysis due to missing baseline data.
Measure: Mean (Standard Deviation); unit: number of hours (self-reported)
Groups:
- Wait-List/Control Treatment With Follow-up (Group B): After the initial 8-week orientation period where Group B will receive 8 weeks of waitlist (limited treatment) control, followed by full access to the "Time for Living & Caring" (TLC) intervention for 8 weeks. They will also receive a 4-week follow-up at Week 20 of the study.
  Time for Living and Caring (TLC): "Time for Living & Caring" (TLC) is an online, self-administered intervention. It includes three types of modules: a "virtual coaching" module (defined as a series or prompts, reminders, and suggestions delivered electronically through an interactive calendar website) that guides caregivers through assessment, goal setting, and goal review activities using an interactive calendar for each planned respite period they have. Supplementary modules provide education and resources such as What is Respite?, Why is Respite Important?, How do I Get (More) Respite?, How do I Use Respite?.
Arm/Group | Treatment With Follow-Up (Group A) | Wait-List/Control Treatment With Follow-up (Group B)
Number analyzed (Participants) | 83 | 80
number of hours (self-reported)
  Pre Intervention | 8.77 (8.89) | 7.81 (11.01)
  Post Intervention | 13.44 (12.64) | 13.11 (10.82)

4. Secondary Outcome: Respite Satisfaction: Count (%) of Participants Who Agreed or Strongly Agreed With the Statement "I am Happy With What I Choose to do During Respite"
Description: Self-report single item measure, assessing partcipants' perceived level of satisfaction with their respite time and time use. Respondents were asked about their level of agreement with the following statement: "I am happy with what I choose to do during my respite time". Responses were recorded on a five-point Likert scale with strongly disagree=1 and strongly agree 5. This variable is dichotomized, showing the count (and percentage) of the sample that responded with "agree" or "stongly agree." This self-report assessment was only collected at baseline (pre-intervention) and at time 16 (post-intervention)
Time Frame: Pre-Intervention (baseline, week 1) and Post-Intervention (week 16) for both Group A and Group B
Population: Three enrolled participants were excluded from this analysis due to missing baseline data.
Measure: Count of Participants; unit: Participants
Groups:
- Waitlist/Control Treatment With Follow-Up (Group B): After the initial 8-week orientation period where Group B will receive 8 weeks of waitlist (limited treatment) control, followed by full access to the "Time for Living & Caring" (TLC) intervention for 8 weeks. They will also receive a 4-week follow-up at Week 20 of the study.
  Time for Living and Caring (TLC): "Time for Living & Caring" (TLC) is an online, self-administered intervention. It includes three types of modules: a "virtual coaching" module (defined as a series or prompts, reminders, and suggestions delivered electronically through an interactive calendar website) that guides caregivers through assessment, goal setting, and goal review activities using an interactive calendar for each planned respite period they have. Supplementary modules provide education and resources such as What is Respite?, Why is Respite Important?, How do I Get (More) Respite?, How do I Use Respite?.
Arm/Group | Treatment With Follow-Up (Group A) | Waitlist/Control Treatment With Follow-Up (Group B)
Number analyzed (Participants) | 83 | 80
Participants
  Pre Intervention (baseline, week 1) | 38 | 34
  Post Intervention (week 16) | 61 | 59

5. Other Pre Specified Outcome: Depressive Symptoms, as Measured by the "PROMIS Depression Scale (Vol 1 Short Form)"
Description: Self-report multi-item index (8-items, additive), with higher scores indicating greater presence and frequency of depressive symptoms; scores are standardized to a distribution of depression-related symptoms on a population-distribution with a mean of 50 and standard deviation of 10 (T-score). Participants self-reported to the following survey questions: "During the past 7 days, I felt worthless, helpless, depressed, hopeless, like a failure, unhappy, that I had nothing to look forward to, that nothing could cheer me up," each assessed with a five-category response (never, rarely, sometimes, often, always). Higher scores indicate a higher level of depressive symptoms.
Time Frame: as for outcome 1
Population: Three enrolled participants were excluded from this analysis due to missing baseline data. If a participant was missing more than 30% of the items (i.e., 2 or more items on the depression questionnaire), the scale score was coded as missing. Under these criteria, the full TLC sample has a calculated score for depression.
Measure: Mean (95% Confidence Interval); unit: T-score
Arm/Group | Treatment With Follow-up (Group A) | Wait-List / Control Treatment With Follow-up (Group B)
Number analyzed (Participants) | 83 | 80
T-score
  T0 - preintervention | 54.34 [52.76 to 55.92] | 53.92 [52.22 to 55.61]
  T4 | 55.81 [54.21 to 57.41] | 55.18 [53.61 to 56.74]
  T8 - mid intervention | 54.68 [52.81 to 56.55] | 54.38 [52.76 to 56.00]
  T12 | 55.73 [53.88 to 57.58] | 53.19 [51.75 to 54.63]
  T16 - post-intervention | 54.75 [52.86 to 56.64] | 52.52 [50.65 to 54.39]
  T20 - follow-up | 56.25 [54.43 to 58.05] | 53.85 [52.08 to 55.62]

ADVERSE EVENTS:
Time Frame: 1 year, 10 months
Description: 1. All-Cause Mortality
  2. Serious Adverse Events
  3. Other (Not Including Serious) Adverse Events
Arm/Group | Treatment With Follow-up (Group A) | Wait-List Control w/Treatment (Group B)
All-Cause Mortality (participants affected / at risk) | 1/83 | 0/83
Serious Adverse Events (participants affected / at risk) | 0/83 | 0/83
Other Adverse Events (participants affected / at risk) | 0/83 | 0/83

LIMITATIONS AND CAVEATS:
NA. The trial was recruited and analyzed as planned.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-09-05): https://cdn.clinicaltrials.gov/large-docs/79/NCT03689179/Prot_SAP_000.pdf
  • Informed Consent Form (2020-07-07): https://cdn.clinicaltrials.gov/large-docs/79/NCT03689179/ICF_001.pdf